CLINICAL TRIAL: NCT04389632
Title: A Phase 1 Study of Sigvotatug Vedotin in Advanced Solid Tumors
Brief Title: A Study of Sigvotatug Vedotin in Advanced Solid Tumors
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Seagen, a wholly owned subsidiary of Pfizer (Industry)
Responsible Party: Sponsor
Organization: Seagen Inc. (Industry)
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: SGNB6A-001; C5751001 (Other: Alias Study Number); 2023-508469-34-00 (Registry Identifier: CTIS (EU))
Record Dates: First submitted 2020-05-12; First posted 2020-05-15 (Actual); Last update posted 2025-12-09 (Actual); Status verified 2025-12

CONDITIONS: Carcinoma, Non-Small Cell Lung; Squamous Cell Carcinoma of Head and Neck; HER2 Negative Breast Neoplasms; Esophageal Squamous Cell Carcinoma; Esophageal Adenocarcinoma; Gastroesophageal Junction Adenocarcinoma; Ovarian Neoplasms; Cutaneous Squamous Cell Cancer; Exocrine Pancreatic Adenocarcinoma; Urinary Bladder Neoplasms; Uterine Cervical Neoplasms; Stomach Neoplasms
Keywords: NSCLC; HNSCC; cSCC; ESCC; EAC; GEJ; HGSOC; Advanced HER2-Negative Breast Cancer; High Grade Serous Ovarian Cancer; Non-Small Cell Lung Cancer; Head and Neck Squamous Cell Cancer; Esophageal Cancer; Bladder Cancer; Cervical Cancer; Gastric Cancer; Seattle Genetics
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung; Squamous Cell Carcinoma of Head and Neck; Esophageal Squamous Cell Carcinoma; Adenocarcinoma Of Esophagus; Ovarian Neoplasms; Urinary Bladder Neoplasms; Uterine Cervical Neoplasms; Stomach Neoplasms; Esophageal Neoplasms | interventions — pembrolizumab; Cisplatin; Carboplatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (5):
- Part A: Dose escalation (Experimental): sigvotatug vedotin monotherapy
  Interventions: Drug: sigvotatug vedotin
- Part B: Dose expansion (Experimental): sigvotatug vedotin monotherapy
  Interventions: Drug: sigvotatug vedotin
- Part C: sigvotatug vedotin combination therapy in NSCLC, HNSCC, ESCC (Experimental): sigvotatug vedotin + pembrolizumab +/- (carboplatin or cisplatin)
  Interventions: Drug: sigvotatug vedotin; Drug: pembrolizumab; Drug: cisplatin; Drug: carboplatin
- Part D: sigvotatug vedotin combination therapy in 1L NSCLC (Experimental): sigvotatug vedotin + pembrolizumab +/- (carboplatin)
  Interventions: Drug: sigvotatug vedotin; Drug: pembrolizumab; Drug: carboplatin
- Part D: sigvotatug vedotin combination therapy in 1L HNSCC (Experimental): sigvotatug vedotin + pembrolizumab +/- (carboplatin or cisplatin)
  Interventions: Drug: sigvotatug vedotin; Drug: pembrolizumab; Drug: cisplatin; Drug: carboplatin

INTERVENTIONS:
Drug: sigvotatug vedotin — Administered into the vein (IV; intravenously)
  Other Names: SGN-B6A; PF-08046047
Drug: pembrolizumab — 200mg every 3 weeks or 400mg every 6 weeks, given by IV
  Other Names: Keytruda
  Arms: Part C: sigvotatug vedotin combination therapy in NSCLC, HNSCC, ESCC; Part D: sigvotatug vedotin combination therapy in 1L HNSCC; Part D: sigvotatug vedotin combination therapy in 1L NSCLC
Drug: cisplatin — 75 mg/m2 every 3 weeks, given by IV
  Arms: Part C: sigvotatug vedotin combination therapy in NSCLC, HNSCC, ESCC; Part D: sigvotatug vedotin combination therapy in 1L HNSCC
Drug: carboplatin — AUC 5 mg/mL per min every 3 weeks, given by IV
  Arms: Part C: sigvotatug vedotin combination therapy in NSCLC, HNSCC, ESCC; Part D: sigvotatug vedotin combination therapy in 1L HNSCC; Part D: sigvotatug vedotin combination therapy in 1L NSCLC

SUMMARY:
This trial will look at a drug called sigvotatug vedotin (SGN-B6A) alone and with pembrolizumab, with or without chemotherapy, to find out whether it is safe for people who have solid tumors. It will study sigvotatug vedotin to find out what its side effects are. A side effect is anything the drug does besides treating cancer. It will also study whether sigvotatug vedotin works to treat solid tumors.

The study will have four parts.

* Part A of the study will find out how much sigvotatug vedotin should be given to participants.
* Part B will use the dose found in Part A to find out how safe sigvotatug vedotin is and if it works to treat solid tumors.
* Part C of the study will find out how safe sigvotatug vedotin is in combination with these other drugs.
* Part D will include people who have not received treatment. This part of the study will find out how safe sigvotatug vedotin is in combination with these other drugs and if these combinations work to treat solid tumors.
* In Parts C and D, participants will receive sigvotatug vedotin with either:

  * Pembrolizumab or,
  * Pembrolizumab and carboplatin, or
  * Pembrolizumab and cisplatin.

ELIGIBILITY:
Inclusion Criteria:

* Disease indication

  * Participants must have histologically or cytologically confirmed metastatic or unresectable solid malignancy within one of the tumor types listed below (dependent on study part).

    * Non-small cell lung cancer (NSCLC)
    * Head and neck squamous cell cancer (HNSCC)
    * Advanced HER2-negative breast cancer
    * Esophageal squamous cell carcinoma (ESCC)
    * Esophageal/Gastro-esophageal junction adenocarcinoma (EAC/GEJ)
    * Cutaneous squamous cell cancer (cSCC)
    * Exocrine pancreatic adenocarcinoma
    * Bladder cancer
    * Cervical cancer
    * Gastric cancer
    * High grade serous ovarian cancer (HGSOC)
  * Part A only: Participants must have disease that is relapsed or refractory or be intolerant to standard-of-care therapies and should have no appropriate standard-of-care therapeutic options.
  * Part B only: Participants must have disease that is relapsed or refractory or be intolerant to standard-of-care therapies. Participants must have received platinum-based therapy and a PD-1/PD-(L)1 inhibitor, if applicable and available.
  * Part C only: For pembrolizumab combination cohorts, participants must be eligible for pembrolizumab per local standard of care. For pembrolizumab with cisplatin or carboplatin, participants must be eligible for both pembrolizumab and the platinum agent per local standard of care. Participants must be treatment naïve for locally advanced or metastatic systemic therapy (prior definitively intended or [neo]adjuvant therapy is allowed).
  * Part D only: Participants must be treatment naïve for locally advanced or metastatic systemic therapy.
* Participants enrolled in the following study parts should have a tumor site accessible for biopsy and agree to biopsy as follows:

  * Disease-specific expansion cohorts (Part B and Part D): A baseline fresh tumor biopsy is required. An archival biopsy collected within 90 days prior to first dose of study drug may be used.
  * Biology expansion cohort: pretreatment biopsy and on-treatment (Cycle 1) biopsy
* An Eastern Cooperative Oncology Group (ECOG) Performance Status of 0 or 1
* Measurable disease per the RECIST v1.1 at baseline

Exclusion Criteria

* History of another malignancy within 3 years before first dose of study drug, or any evidence of residual disease from a previously diagnosed malignancy. Exceptions are malignancies with a negligible risk of metastasis or death.
* Known active central nervous system metastases. Participants with previously treated brain metastases may participate provided they:

  * are clinically stable for at least 4 weeks prior to study entry after brain metastasis treatment,
  * have no new or enlarging brain metastases, and
  * are off of corticosteroids prescribed for symptoms associated with brain metastases for at least 7 days prior to first dose of study drug.
  * In Part D, participants with untreated, asymptomatic CNS metastases smaller than 1 cm may be enrolled without definitive treatment as long as they have no neurological symptoms, no or minimal surrounding edema, and no requirements for corticosteroids.
* Carcinomatous meningitis
* Previous receipt of an MMAE-containing agent or an agent targeting integrin beta-6
* Pre-existing neuropathy Grade 1 or greater per the National Cancer Institute's Common Terminology Criteria for Adverse Events, version 5.0 (NCI CTCAE v5.0) for Parts C and D cohorts with cisplatin or carboplatin; Grade 2 or greater per the NCI CTCAE v5.0 for all other cohorts
* Any uncontrolled Grade 3 or higher (per NCI CTCAE v5.0) viral, bacterial, or fungal infection within 2 weeks prior to the first dose of sigvotatug vedotin.

  * Routine antimicrobial prophylaxis is permitted
* Grade ≥3 pulmonary disease unrelated to underlying malignancy. This includes clinically severe pulmonary function compromise resulting from clinically significant pulmonary illnesses
* Part C and D: Prior therapy with a PD-1 inhibitor, anti-PD-(L)1, or anti PD-L2 agent or with an agent directed to another stimulatory or co-inhibitory T-cell receptor and was discontinued from that treatment due to a Grade 3 or higher immune-mediated adverse event (IMAE).
* History of noninfectious interstitial lung disease (ILD) or pneumonitis that required steroids, current ILD or pneumonitis, or suspected ILD or pneumonitis that cannot be ruled out by imaging at screening
* Known diffusing capacity of the lung for carbon monoxide (DLCO; adjusted for hemoglobin) <50% predicted
* Investigator site staff directly involved in the conduct of the study and their family members, site staff otherwise supervised by the investigator, and sponsor and sponsor delegate employees directly involved in the conduct of the study and their family members.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1006 (Estimated)
Dates: Start 2020-06-08 (Actual); Primary Completion 2027-06-16 (Estimated); Study Completion 2029-03-22 (Estimated)

PRIMARY OUTCOMES:
Number of participants with adverse events (AEs) | Through 30-37 days following last dose of sigvotatug vedotin. For participants receiving pembrolizumab up to 90 days after last dose of pembrolizumab; up to 3 years
  Any untoward medical occurrence in a clinical investigational participant administered a medicinal product and which does not necessarily have a causal relationship with this treatment.
Number of patients with laboratory abnormalities | Through 30-37 days following last dose of sigvotatug vedotin; up to 3 years
Number of participants with dose-limiting toxicities (DLTs) | Through 30-37 days following last dose of sigvotatug vedotin; up to 3 years

SECONDARY OUTCOMES:
Confirmed objective response rate (ORR) per Response Evaluation Criteria in Solid Tumors (RECIST) v1.1 by investigator assessment | Up to approximately 3 years
  The proportion of participants with complete response (CR) or partial response (PR) which is subsequently confirmed as assessed according to RECIST v1.1.
Duration of objective response (DOR) per RECIST v1.1 by investigator assessment | Up to approximately 3 years
  The time from the first documentation of objective response (CR or PR that is subsequently confirmed) to the first documentation of progressive disease (PD) or to death due to any cause
Progression-free survival (PFS) per RECIST v1.1 by investigator assessment | Up to approximately 3 years
  The time from the start of any study treatment to the first documentation of PD, or death due to any cause
Overall survival (OS) | Up to approximately 3 years
  The time from the start of any study treatment to the date of death due to any cause
Area under the concentration-time curve (AUC) | Through 30-37 days following last dose of sigvotatug vedotin; up to 3 years
  Pharmacokinetic (PK) endpoint
Concentration at the end of infusion (Ceoi) | Through 30-37 days following last dose of sigvotatug vedotin; up to 3 years
  PK endpoint
Maximum observed concentration (Cmax) | Through 30-37 days following last dose of sigvotatug vedotin; up to 3 years
  PK endpoint
Time to maximum observed concentration (Tmax) | Through 30-37 days following last dose of sigvotatug vedotin; up to 3 years
  PK endpoint
Trough concentration (Ctrough) | Through 30-37 days following last dose of sigvotatug vedotin; up to 3 years
  PK endpoint
Apparent terminal elimination half-life (t1/2) | Through 30-37 days following last dose of sigvotatug vedotin; up to 3 years
  PK endpoint
Number of participants with antidrug antibodies (ADAs) | Through 30-37 days following last dose of sigvotatug vedotin; up to 3 years

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (149):
- United States (101):
  - Alaska Oncology and Hematology, Anchorage, Alaska
  - Highlands Oncology Group, Fayetteville, Arkansas
  - Highlands Oncology Group, Rogers, Arkansas
  - Highlands Oncology Group, Springdale, Arkansas
  - Providence Medical Foundation, Anaheim, California
  - Providence Medical Foundation, Fullerton, California
  - Providence St. Jude Medical Center Virginia K Crosson and Infusion Center, Fullerton, California
  - Cancer and Blood Research Center, LLC, Los Alamitos, California
  - Cancer and Blood Specialty Clinic, Los Alamitos, California
  - Ronald Reagan UCLA Medical Center, Los Angeles, California
  - The Regents of the University of California, Los Angeles, California
  - UCLA Department of Medicine-Hematology/Oncology, Los Angeles, California
  - UCLA Department of Medicine - Hematology & Oncology, Santa Monica, California
  - Cancer AND Blood Specialty Clinic, Torrance, California
  - American Oncology Partners, PA. a Florida professional service corporation, d/b/a Vista Oncology, Fort Myers, Florida
  - Florida Cancer Specialists & Research Institute, LLC, Fort Myers, Florida
  - Florida cancer Specialists, Fort Myers, Florida
  - Memorial Cancer Institute, Hollywood, Florida
  - Memorial Healthcare System, Hollywood, Florida
  - Florida cancer Specialists, Orlando, Florida
  - Memorial Cancer Institute at Memorial Hospital West, Pembroke Pines, Florida
  - Memorial Hospital West, Pembroke Pines, Florida
  - Ingalls Family Care Center, Calumet City, Illinois
  - UChicago Medicine - River East, Chicago, Illinois
  - The University Of Chicago, Chicago, Illinois
  - University of Chicago Medical Center, Chicago, Illinois
  - UChicago Medicine at Ingalls - Flossmoor, Flossmoor, Illinois
  - UChicago Medicine Ingalls Memorial, Harvey, Illinois
  - University of Chicago Comprehensive Cancer Center at Silver Cross Hospital, New Lenox, Illinois
  - The University of Chicago Medicine Center for Advanced Care Orland Park, Orland Park, Illinois
  - Southern Illinois University - Simmons Cancer Institute, Springfield, Illinois
  - Springfield Clinic Radiology - 800 Building, Springfield, Illinois
  - Springfield Clinic, Springfield, Illinois
  - Springfield Clinic Main Campus, Springfield, Illinois
  - Springfield Clinic Radiology - Main Campus, Springfield, Illinois
  - Springfield Memorial Hospital, Springfield, Illinois
  - UChicago Medicine at Ingalls - Tinley Park, Tinley Park, Illinois
  - UChicago Medicine - Northwest Indiana, Crown Point, Indiana
  - Fort Wayne Medical Oncology and Hematology, Inc, Fort Wayne, Indiana
  - Community Health Network, Inc, Indianapolis, Indiana
  - Community Health Network, Inc., Indianapolis, Indiana
  - Community Health Network Investigational Drug Services, Indianapolis, Indiana
  - Community Health Network, Indianapolis, Indiana
  - The University of Kansas Cancer Center, Investigational Drug Services, Fairway, Kansas
  - The University of Kansas Clinical Research Center, Fairway, Kansas
  - The University of Kansas Hospital, Kansas City, Kansas
  - The University of Kansas Medical Center Medical Office Building, Kansas City, Kansas
  - University of Kansas Hospital Cambridge North Tower A, Kansas City, Kansas
  - University of Kansas Medical Center Research Institute, Kansas City, Kansas
  - The University of Kansas Cancer Center - Indian Creek Campus, Overland Park, Kansas
  - The University of Kansas Cancer Center - Westwood, Westwood, Kansas
  - University of Kansas Cancer Center, Westwood, Kansas
  - Massachusetts General Hospital, Boston, Massachusetts
  - Brigham & Women's Hospital, Boston, Massachusetts
  - Beth Israel Deaconess Medical Center,East Campus Research Pharmacy, Boston, Massachusetts
  - Beth Israel Deaconess Medical Center, Boston, Massachusetts
  - Dana Farber Cancer Institute, Boston, Massachusetts
  - Dana-Farber Cancer Institute - Chestnut Hill, Newton, Massachusetts
  - Allina Health Cancer Institute - Mercy Hospital, Coon Rapids, Minnesota
  - Allina Health Cancer Institute - Abbott Northwestern Hospital, Minneapolis, Minnesota
  - Allina Health Cancer Institute, Saint Paul, Minnesota
  - Comprehensive Cancer Centers of Nevada, Las Vegas, Nevada
  - North Shore Hematology Oncology Associates P.C. DBA New York Cancer and Blood Specialists, Babylon, New York
  - North Shore Hematology Oncology Associates P.C. DBA New York Cancer and Blood Specialists, Brooklyn, New York
  - North Shore Hematology Oncology Associates P.C. DBA New York Cancer and Blood Specialists, New Hyde Park, New York
  - North Shore Hematology Oncology Associates P.C. DBA New York Cancer and Blood Specialists, New York, New York
  - Columbia University Irving Medical Center, New York, New York
  - North Shore Hematology Oncology Associates P.C. DBA New York Cancer and Blood Specialists, Patchogue, New York
  - North Shore Hematology Oncology Associates P.C. DBA New York Cancer and Blood Specialists, Port Jefferson Station, New York
  - North Shore Hematology Oncology Associates P.C. DBA New York Cancer and Blood Specialists, Riverhead, New York
  - North Shore Hematology Oncology Associates P.C. DBA New York Cancer and Blood Specialists, Shirley, New York
  - North Shore Hematology Oncology Associates P.C. DBA New York Cancer and Blood Specialists, The Bronx, New York
  - University Hospitals Cleveland Medical Center, Cleveland, Ohio
  - OU Health University of Oklahoma Medical Center, Oklahoma City, Oklahoma
  - Stephenson Cancer Center (chemo location), Oklahoma City, Oklahoma
  - University of Oklahoma Health Science Center, Oklahoma City, Oklahoma
  - Providence Cancer Institute Franz Clinic, Portland, Oregon
  - Providence Oncology and Hematology Care Clinic - Westside, Portland, Oregon
  - Providence St. Vincent Medical Center- Investigational Drug Services, Portland, Oregon
  - Providence St. Vincent Medical Center, Portland, Oregon
  - Sanford Cancer Center, Sioux Falls, South Dakota
  - Sanford USD Medical Center, Sioux Falls, South Dakota
  - US Oncology Research LLC, Nashville, Tennessee
  - Oncology Consultants, PA, Houston, Texas
  - Oncology Consultants, PA., Houston, Texas
  - The University of Texas M.D. Anderson Cancer Center, Houston, Texas
  - US Oncology Investigational Product Center (IPC), Irving, Texas
  - Houston Medical Imaging, Pearland, Texas
  - South Texas Accelerated Research Therapeutics, LLC, San Antonio, Texas
  - UT Health East Texas HOPE Cancer Center, Tyler, Texas
  - UT Health East Texas Hope Cancer Center, Tyler, Texas
  - Tranquil Clinical Research, Webster, Texas
  - Virginia Cancer Specialists, Fairfax, Virginia
  - Swedish Cancer Institute - Edmonds Campus, Edmonds, Washington
  - Swedish Cancer Institute Edmonds Campus, Edmonds, Washington
  - American Oncology Network Vista Oncology Division-West office, Olympia, Washington
  - American Oncology Network Vista Oncology Division-East office, Olympia, Washington
  - Swedish Cancer Institute, Seattle, Washington
  - Swedish Medical Center, Seattle, Washington
  - Exigent Research, LLC, Tacoma, Washington
  - Northwest Medical Specialities, PLLC, Tacoma, Washington
- France (5):
  - Center Hospitalier Universitaire d' Angers, Angers
  - Institut de Cancérologie de Lorraine, Moselle
  - Centre de Lutte contre le Cancer (CLCC) - Centre Antoine Lacassagne, Nice
  - Centre Hospitalier Universitaire de Poitiers, Poitiers
  - lnstitut Gustave Roussy, Departement d'lnnovation Therapeutique et d'Essais Precoces (DITEP), Villejuif
- South Korea (7):
  - National Cancer Center, Goyang-si, Gyeonggi-do
  - Chungbuk National University Hospital, Cheongju-si
  - Severance Hospital Yonsei University Health System, Seoul
  - Samsung Medical Center, Seoul
  - The Catholic University of Korea, Seoul
  - Seoul National University Boramae Medical Center, Seoul
  - Korea University Guro Hospital, Seoul
- Spain (21):
  - Farmacia Ensayos Hospital HM Universitario Sanchinarro, Madrid, Agrigento
  - Elche General University Hospital, Elche, Alicante
  - Equipo de Farmacia Oncológica- Ensayos Clínicos Servicio de Farmacia Hospital Universitario Marqués, Santander, Cantabria
  - Hospital HM Nou Delfos, Barcelona, Catalonia
  - NEXT Oncology Barcelona - IOB - Hospital Quironsalud Barcelona, Barcelona, OTH
  - Farmacia Ensayos clínicos, Unidad START Barcelona, Barcelona
  - Hospital HM Nou Delfos - START Barcelona, Barcelona
  - Hospital Quiron Salud Barcelona, Barcelona
  - Area general-Planta Baixa | Unitat d'investigacio en terapia Molecular del Cancer "la Caixa", Barcelona
  - Hospital Vall d'Hebron, Barcelona
  - Elche General University Hospital, Elche
  - Hospital Universitario De Jerez, Jerez de la Frontera
  - UGC Farmacia Ensayos clinicos - Hospital Universitario de Jerez, Jerez de la Frontera
  - Hospital Universitario de Jerez, Jerez de la Frontera
  - Fundación de Investigación Hm Hospitales, C.I.F. G-83643841, Madrid
  - Hospital Universitario Ramon y Cajal, Madrid
  - Servicio de Radiologia Hospital Universitario Ramon y Cajal, Madrid
  - Hospital Universitario 12 de Octubre, Madrid
  - Hospital Universitario 12 Octubre, Madrid
  - Hospital HM Sanchinarro, START-Madrid-CIOCC, Madrid
  - Quironsalud Malaga, Málaga
- Switzerland (3):
  - Kantonsspital Graubunden, Chur
  - University Hospital Lausanne CHUV, Lausanne
  - CHUV - Service de pharmacie BH-04, Essais cliniques, Lausanne
- Taiwan (3):
  - Kaohsiung Medical University Hospital, Kaohsiung City, R.o.c.
  - National Taiwan University Hospital, Taipei
  - Taipei Veterans General Hospital., Taipei
- United Kingdom (9):
  - The Royal Marsden Hospital (Surrey), Sutton, Queensland
  - Royal Marsden Hospital, Sutton, Surrey
  - Queen Elizabeth Hospital, Birmingham
  - University Hospitals Birmingham NHS Foundation Trust, Birmingham
  - The Royal Marsden NHS Foundation Trust, London
  - Sarah Cannon Research Institute, London
  - Diagnostic centre, London
  - The Harley Street Clinic, London
  - Radiology, London

IPD SHARING:
Plan to Share IPD: No
Pfizer will provide access to individual de-identified participant data and related study documents (e.g. protocol, Statistical Analysis Plan (SAP), Clinical Study Report (CSR)) upon request from qualified researchers, and subject to certain criteria, conditions, and exceptions. Further details on Pfizer's data sharing criteria and process for requesting access can be found at: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests.

REFERENCES:
- [Derived] Lyon RP, Jonas M, Frantz C, Trueblood ES, Yumul R, Westendorf L, Hale CJ, Stilwell JL, Yeddula N, Snead KM, Kumar V, Patilea-Vrana GI, Klussman K, Ryan MC. SGN-B6A: A New Vedotin Antibody-Drug Conjugate Directed to Integrin Beta-6 for Multiple Carcinoma Indications. Mol Cancer Ther. 2023 Dec 1;22(12):1444-1453. doi: 10.1158/1535-7163.MCT-22-0817. PMID 37619980
- See also: To obtain contact information for a study center near you, click here. — https://pmiform.com/clinical-trial-info-request?StudyID=SGNB6A-001